CLINICAL TRIAL: NCT04376268
Title: Comparison of the Efficacy of Boric Acid Mouthwashes in Different Concentrations in the Lower Third Molar Surgery in the Postoperative Period
Brief Title: Comparison of the Efficacy of Boric Acid Mouthwashes in Different Concentrations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01.08.2018/07
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: postoperative complications; impacted tooth; mouthwash; boric acid; chlorhexidine
MeSH Terms: conditions — Postoperative Complications; Tooth, Impacted | interventions — boric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Chlorhexidine gluconate (Active Comparator): Chlorhexidine is one of the most commonly used medications after tooth extraction. It exhibits a wide spectrum of antiseptic, bactericidal and bacteriostatic effects.
  Interventions: Drug: Chlorhexidine mouthwash
- Chlorhexidine mouthwash with boric acid (0.1%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (0.1%)
- Chlorhexidine mouthwash with boric acid (0.5%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (0.5%)
- Chlorhexidine mouthwash with boric acid (1%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (1%)
- Chlorhexidine mouthwash with boric acid (1.5%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (1.5%)
- Chlorhexidine mouthwash with boric acid (2%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (2%)
- Chlorhexidine mouthwash with boric acid (2.5%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Chlorhexidine mouthwash with boric acid (2.5%)
- Boric acid mouthwash (2%) (Active Comparator): Due to its antibacterial properties, boric acid is effective on gram (+) and gram (-) microorganisms such as candida albicans, streptococcus mutans, staphylococcus aureus, enterococcus faecalis, enterococcus faesium, escherichia coli, klebsiella pneumonia and pseudomonas aeruginosa. With these features, it is used in periodontology, endodontics and restorative therapy as a antiseptic.
  Interventions: Procedure: Boric acid mouthwash (2%)

INTERVENTIONS:
Drug: Chlorhexidine mouthwash — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Other Names: Kloroben Oral Rinse
  Arms: Chlorhexidine gluconate
Procedure: Chlorhexidine mouthwash with boric acid (0.1%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (0.1%)
Procedure: Chlorhexidine mouthwash with boric acid (0.5%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (0.5%)
Procedure: Chlorhexidine mouthwash with boric acid (1%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (1%)
Procedure: Chlorhexidine mouthwash with boric acid (1.5%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (1.5%)
Procedure: Chlorhexidine mouthwash with boric acid (2%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (2%)
Procedure: Chlorhexidine mouthwash with boric acid (2.5%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Chlorhexidine mouthwash with boric acid (2.5%)
Procedure: Boric acid mouthwash (2%) — After anesthesia, the horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under abundant irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with sterile 0.9% saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures. The patients were postoperatively prescribed paracetamol (Parol® 500 mg, Atabay Chemical Industry, Istanbul, Turkey) to use when required with a maximum of 4 doses per day. Patients were instructed to maintain a soft diet, and refrain from mouth washing, brushing and flossing during the first 24 hour. They were also instructed to rinse their mouth with 15 ml of mouthwash for 30 seconds, 3 times a day, and continue until the 7th postoperative day.
  Arms: Boric acid mouthwash (2%)

SUMMARY:
Surgical removal of impacted third molars is one of the most frequent procedures carried out in the oral and maxillofacial surgery clinics. There are a varying range of postoperative complications including pain, edema and swelling. Antibiotics, analgesics and mouthwashes are usually prescribed for the treatment of these complications. Patients undergoing impacted third molar surgery are frequently prescribed chlorhexidine mouthwashes with/without benzydamine hydrochloride. However, there has been a search for alternatives with anti-inflammatory, antibacterial and analgesic properties as part of the oral care routine following surgical removal of impacted third molars. Thus, this multicenter study was aimed to evaluate the effects of chlorhexidine mouthwashes with different boric acid concentrations (%0.1, %0.5, %1, %1.5, %2 and %2.5), and boric acid mouthwash on the postoperative complications and compared with chlorhexidine mouthwash after the removal of impacted wisdom teeth.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease
* having impacted mandibular third molar teeth in a similar position
* absence of allergy to any of the drugs used in the study,
* absence of pregnancy/lactating state,
* no history of any medication use during at least 2 week before the operation.

Exclusion Criteria:

* not regularly coming to the controls,
* not using their medicines regularly
* using any additional medication that may affect the outcome of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative 1st day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Swelling | Postoperatif 1st day
  Facial swelling was assessed using thread and millimeter ruler and five following measurements were taken: Distance I (from angle of the mandible to labial commissure); Distance II (from angle of the mandible to nasal border); Distance III (from angle of the mandible to external corner of the eye); Distance IV (from angle of the mandible to tragus) and Distance V (from angle of the mandible to soft pogonion).
Postoperative Trismus | Postoperative 1st day
  The maximum mouth opening (MMO) was measured in millimeters with a caliper from the incisal edge of the right upper and lower incisor teeth. For evaluation of trismus, the percentage of difference in MMO during postoperative period was calculated by subtracting the preoperative measurement from the postoperative measurement then divided by the preoperative measurement and multiplied by 100.
Postoperative Pain | Postoperative 2nd day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Pain | Postoperative 3rd day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Swelling | Postoperatif 3rd day
  Facial swelling was assessed using thread and millimeter ruler and five following measurements were taken: Distance I (from angle of the mandible to labial commissure); Distance II (from angle of the mandible to nasal border); Distance III (from angle of the mandible to external corner of the eye); Distance IV (from angle of the mandible to tragus) and Distance V (from angle of the mandible to soft pogonion).
Postoperative Trismus | Postoperative 3rd day
  The maximum mouth opening (MMO) was measured in millimeters with a caliper from the incisal edge of the right upper and lower incisor teeth. For evaluation of trismus, the percentage of difference in MMO during postoperative period was calculated by subtracting the preoperative measurement from the postoperative measurement then divided by the preoperative measurement and multiplied by 100.
Postoperative Pain | Postoperative 4th day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Pain | Postoperative 5th day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Pain | Postoperative 6th day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Pain | Postoperative 7th day
  In order to evaluate the postoperative pain, a seven-day scheduled pain diary was given to the patients. To record the level of pain, patients were instructed to rate it on a 10-cm visual analog scales (VAS) was used wherein 0 indicated no pain and 10 indicated the worst pain imaginable.
Postoperative Swelling | Postoperatif 7th day
  Facial swelling was assessed using thread and millimeter ruler and five following measurements were taken: Distance I (from angle of the mandible to labial commissure); Distance II (from angle of the mandible to nasal border); Distance III (from angle of the mandible to external corner of the eye); Distance IV (from angle of the mandible to tragus) and Distance V (from angle of the mandible to soft pogonion).
Postoperative Trismus | Postoperative 7th day
  The maximum mouth opening (MMO) was measured in millimeters with a caliper from the incisal edge of the right upper and lower incisor teeth. For evaluation of trismus, the percentage of difference in MMO during postoperative period was calculated by subtracting the preoperative measurement from the postoperative measurement then divided by the preoperative measurement and multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No